CLINICAL TRIAL: NCT06329791
Title: A Phase 3, Multicenter, Vehicle-controlled, Randomized Study to Evaluate the Efficacy, Safety, and Tolerability of AZR-MD-001 in Patients with Abnormal Meibomian Gland Function and Associated Symptoms of Dry Eye Disease (DED)
Brief Title: A Phase 3 Study to Evaluate AZR-MD-001 in Patients with Abnormal Meibomian Gland Function and Dry Eye Disease (DED)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azura Ophthalmics (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AZ202401
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-06

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AZR-MD-001 (Experimental): AZR-MD-001 sterile ophthalmic ointment 0.5% to be administered twice weekly at bedtime.
  Interventions: Drug: AZR-MD-001
- Vehicle (Placebo Comparator): AZR-MD-001 Vehicle to be administered twice weekly at bedtime.
  Interventions: Other: Vehicle

INTERVENTIONS:
Drug: AZR-MD-001 — AZR-MD-001 sterile ophthalmic ointment 0.5%
  Other Names: AZR-MD-001 ophthalmic ointment 0.5%
  Arms: AZR-MD-001
Other: Vehicle — AZR-MD-001 Vehicle
  Other Names: AZR-MD-001 Vehicle
  Arms: Vehicle

SUMMARY:
This study is a multicenter, double-masked, vehicle-controlled, randomized, parallel group study designed to evaluate the treatment of abnormal meibomian gland function and associated symptoms of DED using either AZR-MD-001 0.5% ophthalmic ointment or its vehicle. Study drug (either AZR-MD-001 or vehicle) will be dosed twice-weekly at bedtime for up to 12 months.

DETAILED DESCRIPTION:
This study is designed to evaluate the treatment of abnormal meibomian gland function and associated symptoms of DED using either AZR-MD-001 0.5% ophthalmic ointment or its vehicle. Study drug (either AZR-MD-001 or vehicle) will be dosed twice-weekly at bedtime for up to 12 months.

Following a Screening qualification period, all patients diagnosed with abnormal meibomian gland function and associated symptoms of DED, and meeting the inclusion/exclusion criteria, will be randomized centrally, to treatment in a 1:1 ratio.

Study follow-up visits will be conducted on Day 14, Month 1.5, Month 3, Month 4.5, Month 6, Month 9, and Month 12. Patients will exit the study approximately 13 months after the Baseline visit. Any ongoing treatment-emergent adverse events (TEAEs) will be followed for an additional 30 days following the Month 12 visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older at Screening.
* Evidence of active Evaporative DED at Screening and Baseline.
* Evidence of meibomian gland obstruction in both eyes at Screening and Baseline.

Exclusion Criteria:

* Ocular disease (except for Meibomian Gland Dysfunction (MGD) and DED/keratoconjunctivitis sicca) or systemic disease determined to be uncontrolled by the investigator.
* Patient has glaucoma, ocular hypertension, or an intraocular pressure (IOP) of ≥24 mm Hg in either eye at Screening.
* Recent (within the past 3 months of Screening) ocular surgery, trauma, herpes, or recurrent inflammation.
* Unwilling to abstain from the use of systemic or topical treatments for MGD or dry eye for the study duration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Meibomian Glands Yielding Liquid Secretion | Month 3
  Meibomian Glands Yielding Liquid Secretion (MGYLS) measures the number of meibomian glands (0 - 15) secreting liquid
Change from baseline in Total Ocular Surface Disease Index Score | Month 3
  The Total Ocular Surface Disease Index Score (OSDI) provides a score from 0 (normal) to 100 (abnormal)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Bosworth, PhD, Study Director — Azura Ophthalmics
Locations (16):
- United States (16):
  - Arizona Eye Center, Chandler, Arizona
  - Global Research Management, Inc, Glendale, California
  - Eye Research Foundation, Newport Beach, California
  - NVISION Clinical Research, Torrance, California
  - Wyse Eyecare, Northbrook, Illinois
  - Pankratz Eye Institute, Columbus, Indiana
  - The Eye Care Institute/Butchertown Clinical Trials, Louisville, Kentucky
  - Ophthalmology Associates, St Louis, Missouri
  - NC Eye Associates, Apex, North Carolina
  - Oculus Research, Inc., Garner, North Carolina
  - CORE, Shelby, North Carolina
  - Scott & Christie and Associates, PC, Cranberry Township, Pennsylvania
  - Advancing Vision Research (AVR) - Goodlettsville, Goodlettsville, Tennessee
  - Total Eye Care, Memphis, Tennessee
  - Advancing Vision Research (AVR) - Smyrna, Smyrna, Tennessee
  - Piedmont Eye Center, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No